CLINICAL TRIAL: NCT00197990
Title: Expectations, Satisfaction and Quality of Life in Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 22078; Arthritis Foundation-NY Chapt
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Hip Osteoarthritis; Arthroplasty, Replacement, Hip
Keywords: total hip arthroplasty; expectations; satisfaction; quality of life
MeSH Terms: conditions — Osteoarthritis, Hip; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goals of this study are to identify predictors of improvement in quality of life and satisfaction with total hip arthroplasty three to five years after surgery.

DETAILED DESCRIPTION:
The goals of this study are to identify predictors of improvement in quality of life and satisfaction with total hip arthroplasty three to five years after surgery. Predictors that will be considered are variables that were obtained prospectively and systematically at the time of surgery, including demographic characteristics, functional status, expectations, perioperative complications, and comorbidity. At the follow-up functional status and patient satisfaction will be measured, as well as fulfillment of expectations and predispositional factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for this study if they are part of an assembled cohort of patients who underwent primary unilateral or bilateral total hip arthroplasty in 1998-2000 at the Hospital for Special Surgery.

Exclusion Criteria:

* Patients will be excluded if they are unable to be interviewed, refuse to participate, or are deceased.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had total hip arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2003-07; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Fulfillment of expectations

SECONDARY OUTCOMES:
Satisfaction with THA

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Mancuso, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Mancuso CA, Sculco TP, Salvati EA. Patients with poor preoperative functional status have high expectations of total hip arthroplasty. J Arthroplasty. 2003 Oct;18(7):872-8. doi: 10.1016/s0883-5403(03)00276-6. PMID 14566742
- [Background] Mancuso CA, Salvati EA, Johanson NA, Peterson MG, Charlson ME. Patients' expectations and satisfaction with total hip arthroplasty. J Arthroplasty. 1997 Jun;12(4):387-96. doi: 10.1016/s0883-5403(97)90194-7. PMID 9195314
- [Background] Mancuso CA, Ranawat CS, Esdaile JM, Johanson NA, Charlson ME. Indications for total hip and total knee arthroplasties. Results of orthopaedic surveys. J Arthroplasty. 1996 Jan;11(1):34-46. doi: 10.1016/s0883-5403(96)80159-8. PMID 8676117
- [Background] Blake VA, Allegrante JP, Robbins L, Mancuso CA, Peterson MG, Esdaile JM, Paget SA, Charlson ME. Racial differences in social network experience and perceptions of benefit of arthritis treatments among New York City Medicare beneficiaries with self-reported hip and knee pain. Arthritis Rheum. 2002 Aug;47(4):366-71. doi: 10.1002/art.10538. PMID 12209481
- [Background] Peterson MG, Hollenberg JP, Szatrowski TP, Johanson NA, Mancuso CA, Charlson ME. Geographic variations in the rates of elective total hip and knee arthroplasties among Medicare beneficiaries in the United States. J Bone Joint Surg Am. 1992 Dec;74(10):1530-9. PMID 1469013
- [Result] Mancuso CA, Jout J, Salvati EA, Sculco TP. Fulfillment of patients' expectations for total hip arthroplasty. J Bone Joint Surg Am. 2009 Sep;91(9):2073-8. doi: 10.2106/JBJS.H.01802. PMID 19723982